CLINICAL TRIAL: NCT05734287
Title: Polycystic Ovaries in Young Girls Presenting With Hyperandrogenism
Brief Title: The Frequency of Polycystic Ovary Syndrome Among Young Reproductive Females Presenting With Hyperandrogenism: a Mixed Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Other Study IDs: 123456
Record Dates: First submitted 2023-02-06; First posted 2023-02-17 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: clinical, biophysical and biochemical assessment of young females with clinical hyperandrogenism — To assess clinical, biophysical and biochemical criteria of young females with clinical hyperandrogenism as a search for PCOS

SUMMARY:
This mixed cohort study will test the frequency of PCOS among young females presenting with one of the clinical hyperandrogenism criteria: acne, hirsutism and/or hair loss. Diagnosis will be based on the recent PCOS clinical, biochemical and biophysical criteria recently published " International evidence-based guideline for the assessment and management of polycystic ovary syndrome (PCOS) 2018".

DETAILED DESCRIPTION:
Irregular menstrual cycles are defined as:

* normal in the first year post menarche as part of the pubertal transition
* > 1 to < 3 years post menarche: < 21 or > 45 days
* > 3 years post menarche to perimenopause: < 21 or > 35 days or < 8 cycles per year
* > 1 year post menarche > 90 days for any one cycle
* Primary amenorrhea by age 15 or > 3 years post thelarche (breast development) When irregular menstrual cycles are present a diagnosis of PCOS should be considered.

Biochemical hyperandrogenism: Calculated free testosterone, free androgen index or calculated bioavailable testosterone. Androstenedione and dehydroepiandrosterone sulfate (DHEAS) could be considered if total or free testosterone are not elevated. (ELIZA or radioimmunoassay).

A comprehensive history and physical examination should be completed for symptoms and signs of clinical hyperandrogenism, including acne, alopecia and hirsutism and, in adolescents, severe acne and hirsutism using the modified Ferriman Gallwey score (mFG). Transvaginal (transabdominal if virgins) Ultrasound and polycystic ovarian morphology: Ultrasound should not be used for the diagnosis of PCOS in those with a gynaecological age of < 8 years (< 8 years after menarche), due to the high incidence of multi-follicular ovaries in this life stage. Transabdominal ultrasound reporting is best focused on ovarian volume with a threshold of ≥ 10ml. Endovaginal U/S should show a follicle number per ovary of ≥ 20 and/or an ovarian volume ≥ 10ml, ensuring no corpora lutea, cysts or dominant follicles are present.

ELIGIBILITY:
Inclusion Criteria:

* Clinical hyperandrogenism

Exclusion Criteria:

* Age less than 15 or more than 35 years.

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Females with clinical hyperandrogenism.
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The frequency of polycystic ovary syndrome among young reproductive females presenting with hyperandrogenism: a mixed cohort study | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Atif Dervis, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
Protocol
Supporting Information: Study Protocol
Time Frame: 3 months